**Unique Protocol ID: No.2024018** 

Official Title: Transcranial electrical stimulation combined with interim testing promotes temporal memory in patients with schizophrenia

**Document Title: Informed Consent** 

Date of the Document: 2024/07/15

| Informed Consent | |
|---|---|
| Clinical Research Programs | : Transcranial electrical stimulation combined with interim testing |
| promot | es temporal memory in patients with schizophrenia |
| Project Organizer: | Northwest Normal University |
| Project Collaborators: | The Third People's Hospital of Lanzhou |
| Statement of Consent | |
| Dear Patient: | |
| č | I to participate in a study on memory. The study protocol has been<br>the Ethics Committee of Northwest Normal University and the<br>nzhou City for the study. |
| | you agree to the following: |
| <ul><li>I have read and unde</li></ul> | erstood the protocol in its entirety. |
| • The experimenter ha | s answered any questions I may have about this experiment. |
| • I can ask to stop the | he experiment at any time if I feel any discomfort during the |
| experiment. | |
| I have been informe | d that all experimental content will be kept confidential and will |
| not be made public in any wa | y that identifies an individual, unless required by law. |
| Finally, I have voluntaril | ly decided to participate in this study. |
| | Patient's signature: |
| I confirm that the detain powers and possible benefits | ls of this trial have been explained to the patient, including its and risks. |
| | Signature of the doctor: |